CLINICAL TRIAL: NCT03440905
Title: Proxy-Reported Symptoms and Quality of Life Survey in Zellweger Spectrum Disorders
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Montclair State University (Other); University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: STAIR 7010
Record Dates: First submitted 2018-02-13; First posted 2018-02-22 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Zellweger Spectrum
MeSH Terms: conditions — Zellweger Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to characterize the symptoms of Zellweger Spectrum Disorder (ZSD) and related peroxisome disorders, and to assess the quality of life of family caregivers (parents, stepparents, legal guardians) of patients diagnosed with ZSD or a related peroxisome disorder. All family caregivers of patients enrolled in the Rare Diseases Clinical Research Network (RDCRN) Contact Registry who are diagnosed with ZSD or a related peroxisome disorder will be invited via email to participate in this study.

DETAILED DESCRIPTION:
A total of three online surveys will be provided to each family caregiver that fits the inclusion criteria and is enrolled in the RDCRN STAIR Contact Registry. All three surveys should take approximately 60 minutes total to complete.

The first survey included is the ZSD Symptom Inventory, which is comprised of both multiple choice and open-ended responses. The survey asks family caregivers multiple questions regarding their child's mobility, balance, vision, and hearing status, as well as when they were diagnosed, test results, and past and present symptoms. This survey was adapted from an instrument that was developed by a physician-researcher in the field of ZSD to correlate caregiver-reported symptoms of ZSD to metabolic markers of ZSD (Wangler et al. Manuscript submitted, Pediatrics). For the purpose of this study, the survey was expanded to include domains that were determined based on existing literature on clinical symptoms of ZSD as well as input from both expert clinicians in the field and parents of children diagnosed with ZSD. Both clinicians and parents were in agreement that the questions included in the survey were comprehensive, appropriate and relevant for ZSD. Additionally, pilot testing of this survey to 34 family ZSD caregivers (26 parents of living children, 8 parents of deceased children) provided feedback on increasing the answer choice options for the survey, and adding more open-ended questions. This survey will take an estimated 40 minutes to complete. Family caregivers of living and deceased children will take this survey, and the tense and recall language will be modified to accommodate each of these experiences.

The second survey is the Pediatric Inventory for Parents (PIP) Survey. It includes 42 Likert-scale questions; for each question asked, two sets of responses need to be completed, including responses to "how often" and "how difficult" each topic is for the patient or family caregiver over a given period of time. The PIP measures four domains including communication, medical care, emotional distress, and role function. This instrument has been validated to assess caregiver burden in multiple pediatric chronic illnesses, including type I diabetes, inflammatory bowel disease, and multiple congenital disorders including mitochondrial disease. Although this is validated in parents of living children with pediatric illnesses, the investigators will also be administering a modified PIP to ZSD family caregivers of deceased children, asking them to recall their experience over the last 12 months of their child's life. The PIP takes an estimated 10 minutes to complete.

The third survey is the Family Quality of Life (FQOL) Survey. It includes 25 Likert-scale questions, regarding how parents/primary caregivers feel about his or her life together as a family over a given period of time. The FQOL measures 5 domains including family interaction, parenting, emotional well-being, physical/material well-being, and disability-related support, and has been validated for use in families of children with disabilities. Although this is validated in parents of living children with disabilities, the investigators will also be administering a modified FQOL to ZSD family caregivers of deceased children, asking them to recall their experience over the last 12 months of their child's life. The FQOL takes less than 10 minutes to complete.

The PIP and the FQOL were chosen for this study as they are validated tools for assessing quality of life in caregivers for chronic pediatric illnesses (PIP) and for children with disabilities (FQOL). Although many of these diseases that have been used for validation of these instruments are clinically distinct from ZSD, we expect there to be similarities in the caregiver experience between ZSD and these diseases in the domains of communication, medical care, emotional distress, family interaction, parenting, physical well-being and disability-related support. As a rare disease, the relatively low prevalence of the ZSD and likely decreased awareness may affect certain domains differently than the more common diseases that have been studied using these tools. Nevertheless, the PIP is one of the most commonly used survey tools for caregiver quality of life in chronic pediatric illnesses [8]. The FQOL is currently one of the only tools for assessing quality of life in caregivers for children with disabilities. This is one of the first studies assessing quality of life in families affected by ZSD; the information gained from this study can be used to help shape future quality of life studies in ZSD and other rare disease populations as well as ultimately be used to determine the impact of the disease and emerging treatments.

All participants will have 2 months from the time that they complete the consent form to complete all 3 surveys. Recruitment for the study will close 6 months from the survey launch date.

The survey data will be stored by the RDCRN's Data Management and Coordinating Center (DMCC) at the University of South Florida (USF). The RDCRN Contact Registry collects the names, phone numbers, and addresses of registrants. All data collected will be sent to the database of Genotypes and Phenotypes (dbGaP) to be stored indefinitely.

ELIGIBILITY:
Inclusion Criteria:

* Family caregiver (parents, stepparents, legal guardians) of child (living or deceased) diagnosed with ZSD, acyl CoA oxidase (ACOX) deficiency or D-bifunctional protein deficiency (DBPD)
* Family caregiver is able to complete surveys

Exclusion Criteria:

* Inability of family caregiver to provide informed consent and complete survey
* Parents/primary caregivers of children who have not been diagnosed with ZSD, acyl CoA oxidase deficiency and D-bifunctional protein deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Family caregivers (parents, stepparents, legal guardians) of patients (living or deceased) with ZSD or related peroxisome disorder diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Characterization of Symptoms | 6 months from the study start date
  To characterize the symptoms of Zellweger spectrum disorder (ZSD) and related peroxisome disorders through family caregiver-reported measures using a customized survey tool.

SECONDARY OUTCOMES:
Quality of Life Assessment | 6 months from the study start date
  To assess quality of life for family caregivers of children with ZSD and related peroxisome disorders through the domains of communication, medical care, emotional distress and well-being, role function, family interaction, parenting, and disability-related support, using the validated Pediatric Inventory for Parents (PIP).
Quality of Life Assessment | 6 months from the study start date
  To assess quality of life for family caregivers of children with ZSD and related peroxisome disorders through the domains of communication, medical care, emotional distress and well-being, role function, family interaction, parenting, and disability-related support, using the FQOL Survey.

OTHER OUTCOMES:
Quality of Life Caregiver-reported Comparison | 6 months from the study start date
  To compare family caregiver-reported quality of life between male and female family caregivers of children with ZSD and related peroxisome disorders through the domains of communication, medical care, emotional distress and well-being, role function, family interaction, parenting, and disability-related support, using the validated Pediatric Inventory for Parents (PIP).
Quality of Life Caregiver-reported Comparison | 6 months from the study start date
  To compare family caregiver-reported quality of life between male and female family caregivers of children with ZSD and related peroxisome disorders through the domains of communication, medical care, emotional distress and well-being, role function, family interaction, parenting, and disability-related support, using the FQOL Survey.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States

REFERENCES:
- [Background] Braverman NE, Raymond GV, Rizzo WB, Moser AB, Wilkinson ME, Stone EM, Steinberg SJ, Wangler MF, Rush ET, Hacia JG, Bose M. Peroxisome biogenesis disorders in the Zellweger spectrum: An overview of current diagnosis, clinical manifestations, and treatment guidelines. Mol Genet Metab. 2016 Mar;117(3):313-21. doi: 10.1016/j.ymgme.2015.12.009. Epub 2015 Dec 23. PMID 26750748
- [Background] Klouwer FC, Berendse K, Ferdinandusse S, Wanders RJ, Engelen M, Poll-The BT. Zellweger spectrum disorders: clinical overview and management approach. Orphanet J Rare Dis. 2015 Dec 1;10:151. doi: 10.1186/s13023-015-0368-9. PMID 26627182
- [Background] Streisand R, Braniecki S, Tercyak KP, Kazak AE. Childhood illness-related parenting stress: the pediatric inventory for parents. J Pediatr Psychol. 2001 Apr-May;26(3):155-62. doi: 10.1093/jpepsy/26.3.155. PMID 11259517
- [Background] Senger BA, Ward LD, Barbosa-Leiker C, Bindler RC. The Parent Experience of Caring for a Child with Mitochondrial Disease. J Pediatr Nurs. 2016 Jan-Feb;31(1):32-41. doi: 10.1016/j.pedn.2015.08.007. Epub 2015 Oct 9. PMID 26453412
- [Background] Gray WN, Graef DM, Schuman SS, Janicke DM, Hommel KA. Parenting stress in pediatric IBD: relations with child psychopathology, family functioning, and disease severity. J Dev Behav Pediatr. 2013 May;34(4):237-44. doi: 10.1097/DBP.0b013e318290568a. PMID 23669870
- [Background] Caris EC, Dempster N, Wernovsky G, Butz C, Neely T, Allen R, Stewart J, Miller-Tate H, Fonseca R, Texter K, Nicholson L, Cua CL. Anxiety Scores in Caregivers of Children with Hypoplastic Left Heart Syndrome. Congenit Heart Dis. 2016 Dec;11(6):727-732. doi: 10.1111/chd.12387. Epub 2016 Jun 20. PMID 27320439
- [Background] Park J, Hoffman L, Marquis J, Turnbull AP, Poston D, Mannan H, Wang M, Nelson LL. Toward assessing family outcomes of service delivery: validation of a family quality of life survey. J Intellect Disabil Res. 2003 May-Jun;47(Pt 4-5):367-84. doi: 10.1046/j.1365-2788.2003.00497.x. PMID 12787167
- [Background] Cousino MK, Hazen RA. Parenting stress among caregivers of children with chronic illness: a systematic review. J Pediatr Psychol. 2013 Sep;38(8):809-28. doi: 10.1093/jpepsy/jst049. Epub 2013 Jul 10. PMID 23843630
- [Background] Theil AC, Schutgens RB, Wanders RJ, Heymans HS. Clinical recognition of patients affected by a peroxisomal disorder: a retrospective study in 40 patients. Eur J Pediatr. 1992 Feb;151(2):117-20. doi: 10.1007/BF01958955. PMID 1371465
- [Background] Nasrallah F, Zidi W, Feki M, Kacem S, Tebib N, Kaabachi N. Biochemical and clinical profiles of 52 Tunisian patients affected by Zellweger syndrome. Pediatr Neonatol. 2017 Dec;58(6):484-489. doi: 10.1016/j.pedneo.2016.08.011. Epub 2017 Feb 17. PMID 28330580
- [Background] Poll-The BT, Gootjes J, Duran M, De Klerk JB, Wenniger-Prick LJ, Admiraal RJ, Waterham HR, Wanders RJ, Barth PG. Peroxisome biogenesis disorders with prolonged survival: phenotypic expression in a cohort of 31 patients. Am J Med Genet A. 2004 May 1;126A(4):333-8. doi: 10.1002/ajmg.a.20664. PMID 15098231
- [Background] Johnston BC, Miller PA, Agarwal A, Mulla S, Khokhar R, De Oliveira K, Hitchcock CL, Sadeghirad B, Mohiuddin M, Sekercioglu N, Seweryn M, Koperny M, Bala MM, Adams-Webber T, Granados A, Hamed A, Crawford MW, van der Ploeg AT, Guyatt GH. Limited responsiveness related to the minimal important difference of patient-reported outcomes in rare diseases. J Clin Epidemiol. 2016 Nov;79:10-21. doi: 10.1016/j.jclinepi.2016.06.010. Epub 2016 Jul 2. PMID 27381737
- [Background] Dinour LM, Pope GA, Bai YK. Breast milk pumping beliefs, supports, and barriers on a university campus. J Hum Lact. 2015 Feb;31(1):156-65. doi: 10.1177/0890334414557522. Epub 2014 Nov 11. PMID 25389127
- [Background] Dinour LM, Pole A. Potato Chips, Cookies, and Candy Oh My! Public Commentary on Proposed Rules Regulating Competitive Foods. Health Educ Behav. 2017 Dec;44(6):867-875. doi: 10.1177/1090198117699509. Epub 2017 Apr 6. PMID 28382838
- [Background] Dinour LM. Conflict and compromise in public health policy: analysis of changes made to five competitive food legislative proposals prior to adoption. Health Educ Behav. 2015 Apr;42(1 Suppl):76S-86S. doi: 10.1177/1090198114568303. PMID 25829121